CLINICAL TRIAL: NCT01669629
Title: Comparison of Two Daily Disposable Contact Lenses Over 1-week of Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CR-005199
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delefilcon A/ Etafilcon A (Experimental): 6-10 days of delefilcon A soft contact lens wear first, then 6-10 days of etafilcon A soft contact lens wear
  Interventions: Device: delefilcon A; Device: etafilcon A
- Etafilcon A / Delefilcon A (Experimental): 6-10 days of etafilcon A soft contact lens wear first then 6-10 days of delefilcon A soft contact lens wear
  Interventions: Device: delefilcon A; Device: etafilcon A

INTERVENTIONS:
Device: delefilcon A — Daily wear soft contact lens for bilateral distance vision correction use.
Device: etafilcon A — Daily wear soft contact lens for bilateral distance vision correction use.

SUMMARY:
This is a one week 2x2 crossover study comparing delefilcon A with etafilcon A, with a primary hypothesis of comparing the handling of each lens. Additional secondary markers are measured looking at subjective comfort and vision of the lenses.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be between 18 and 45 years of age (inclusive) with no presbyopic add.
* The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form. This should be recorded on the Case Report Form (CRF).
* The subject must be willing to wear the study lenses for at least 8 hours per day, 7 days per week.
* The subject must be a current successful soft contact lens wearer in both eyes
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* The subject's subjective refraction must result in a vertex corrected spherical contact lens prescription in the range of -1.00D to -6.00D in each eye.
* The subject's refractive astigmatism must be less than or equal to 0.75D in both eyes.
* The subject must have best corrected visual acuity of 20/30 (6/9) or better in each eye.
* The subject must require a visual correction in both eyes (no monofit or monovision allowed).
* The subject must have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:

  1. No amblyopia.
  2. No evidence of lid abnormality or infection (including blepharitis/meibomitis).
  3. No conjunctival abnormality or infection.
  4. No clinically significant slit lamp findings (i.e. stromal edema, vascularization, infiltrates or abnormal opacities).
  5. No other active ocular disease.

Exclusion Criteria:

* Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
* Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear.
* Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (Grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation.
* No extended wear in the last 3 months.
* Diabetes.
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immunosuppressive disease (e.g. HIV).
* Employee or family member of the staff of the investigational site.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Little Rock, Arkansas
  - Bridgeport, Connecticut
  - Tampa, Florida
  - Blue Springs, Missouri
  - Vestal, New York
  - Raleigh, North Carolina
  - Kittanning, Pennsylvania
  - Warwick, Rhode Island
  - Chamberlain, South Dakota
  - Bartlett, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 183 subjects enrolled with 183 subjects randomized.
Groups:
- Delefilcon A \ Etafilcon A: 6-10 days of delefilcon A soft contact lens wear first then 6-10 days of etafilcon A soft contact lens wear
  delefilcon A: Daily wear soft contact lens for bilateral distance vision correction use.
  etafilcon A: Daily wear soft contact lens for bilateral distance vision correction use.
- Etafilcon A \ Delefilcon A: 6-10 days of etafilcon A soft contact lens wear first then 6-10 days of delefilcon A soft contact lens wear
  delefilcon A: Daily wear soft contact lens for bilateral distance vision correction use.
  etafilcon A: Daily wear soft contact lens for bilateral distance vision correction use.
Period: Period 1
Arm/Group | Delefilcon A \ Etafilcon A | Etafilcon A \ Delefilcon A
Started | 92 | 91
Completed | 91 | 89
Not Completed | 1 | 2
Not completed — protocol deviation | 1 | 2
Period: Period 2
Arm/Group | Delefilcon A \ Etafilcon A | Etafilcon A \ Delefilcon A
Started | 91 | 89
Completed | 91 | 89
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects.
Groups:
- All Subjects: All subjects who were enrolled in the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.61 (7.061)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125
  Male | 58
Region of Enrollment [Number; unit: participants]
  United States | 183

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Ease of Removal
Description: Measured on a 5 point-scale of excellence (excellent, very good, good, fair and poor) per a participant. Outcome is reported as aggregate number of subjects who reported Excellent/Very Good at their 1-week visit.
Time Frame: 6-10 Days
Population: Subjects analyzed were those who enrolled, randomized, and completed the study per protocol.
Measure: Number; unit: percentage of participants
Groups:
- Delefilcon A: Subjects that received the delefilcon A lens in either the first or second period of the study.
- Etafilcon A: Subjects that received the etafilcon A lens in either the first or second period of the study.
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 180 | 180
percentage of participants | 47.2 | 75.6

2. Secondary Outcome: Subject Reported Overall Comfort
Description: Measured on a 5 point-scale of excellence (excellent, very good, good, fair and poor) per a participant. Summary is reported as an aggregate of Excellent/Very Good at their 1-week visit.
Time Frame: 6-10 Days
Measure: Number; unit: percentage of participants
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 180 | 180
percentage of participants | 71.1 | 61.1

3. Secondary Outcome: Subject Reported Overall Vision
Description: Measured on a 5 point-scale of excellence (excellent, very good, good, fair and poor) per a participant using an aggregate summary of excellent/very good at their 1-week visit.
Time Frame: 6-10 Days
Measure: Number; unit: percentage of participants
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 180 | 180
percentage of participants | 76.1 | 72.2

4. Secondary Outcome: Binocular Snellen Visual Acuity
Description: Snellen visual acuity percentage of eyes with a visual acuity of eyesight testing at a 20/20 level or better by eye.
Time Frame: 6-10 Days
Population: Subjects are those who were enrolled, randomized, and completed the study per protocol. Number of subjects is total in sample due to stratification by device and binocular measurement setting only.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 180 | 180
Number analyzed (Eyes) | 360 | 360
percentage of eyes | 95.0 | 94.7

5. Secondary Outcome: Overall Corneal Staining
Description: Proportion of subjects that have corneal staining on the 0-4 the NEI/Industry Workshop guidelines scale, measured by eye.
  Grade 1 or higher is reported as a percentage of total eyes.
Time Frame: 6-10 Days
Population: Subjects are those who were enrolled, randomized, and completed the study per protocol. Percentage of eyes.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Delefilcon A | Etafilcon A
Number analyzed (Participants) | 180 | 180
Number analyzed (eyes) | 360 | 360
percentage of eyes | 19.4 | 11.9

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 2 weeks.
Groups:
- Etafilcon A: Subjects that received the delefilcon A lens in either the first or second period of the study.
Arm/Group | Delefilcon A | Etafilcon A
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days